CLINICAL TRIAL: NCT03626155
Title: Does Exercise Timing Affect Glucose Levels in People With Diabetes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Normand Boule, Professor, University of Alberta
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00078578
Record Dates: First submitted 2018-07-09; First posted 2018-08-10 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Walking; type 2 diabetes; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Seated Control (Experimental)
  Interventions: Behavioral: Seated Control
- Morning Exercise (walking) (Experimental)
  Interventions: Behavioral: Walking
- Afternoon Exercise (walking) (Experimental)
  Interventions: Behavioral: Walking
- Evening Exercise (walking) (Experimental)
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Walking will last 50 minutes and will be at 5.0 km/h and at 0.5% incline
  Arms: Afternoon Exercise (walking); Evening Exercise (walking); Morning Exercise (walking)
Behavioral: Seated Control — Participants will be asked to sit quietly and read during a 50 minute control period
  Arms: Seated Control

SUMMARY:
It is not clear if there is an optimal time for exercise to improve blood glucose profiles in people with type 2 diabetes. The goal of this study is to compare post meal and 24-hour glucose levels in 4 different conditions: i-seated control, ii-fasted state exercise, iii-30 minutes post meal exercise, and iv- 3-4-hour post meal exercise. The primary outcome of this study is glucose control assessed over 24 hours using continuous glucose monitoring.

DETAILED DESCRIPTION:
Purpose:To compare the effects of a single bout of walking conducted at different times of the day on 24-hour glucose profiles in individuals with type 2 diabetes. In addition to a control (no exercise) conditions, a bout of walking will be completed in the following 3 conditions i. in the fasted state, before breakfast, ii. 3-4 hours after lunch, and iii. 30 minutes after dinner.

Background: Recently, we developed the Exercise-Physical Activity and Diabetes Glucose Monitoring (E-PAraDiGM), which was tested at 8 different sites across Canada (ClinicalTrials.gov Identifier: NCT02834689). The original E-PAraDiGM protocol found no significant difference in 24-hour glucose levels between the exercise and seated control condition (publication in preparation). One the of the potential reasons for this could be the timing of exercise in relation to meals. There is no clear consensus as to the optimal time for exercise for individuals with type 2 diabetes. The goal of this study is to expand on the original E-PAraDiGM study by adding fasted state exercise and 30 minute postprandial exercise to the original 2 conditions (3-4 hours after lunch and seated control).

Research Design: The complete protocol will take place over two separate 6-day periods for each participant, which includes 50 minutes of exercise done in the following 4 conditions i. in the fasted state, before breakfast, ii. 3-4hrs after lunch, iii. 30 minutes after dinner, and iv. seated control. Each participant will complete each condition according to a randomized, crossover design.

Participants: Twelve individuals with T2D will be recruited at the University of Alberta. Participants will be between the ages of 30-90 years and will have been diagnosed with T2D for more than 6 months. They will also have no contraindications to exercise, no previous myocardial infarction, strokes, or coronary artery disease. Participants will not be treated with insulin or corticosteroids and they will have had no changes in diabetes medications in the last 3 months. Furthermore, participants will have no significant changes in body weight (>5%) in the last 3 months. Their blood pressure will be below 160/100 mmHg and their resting heart rate will be below 100 beats per minute.

Baseline Assessment: An initial visit will be used to perform screening, obtain written informed consent, and collect baseline data, including: anthropometry (e.g., height, weight, waist/hip circumference), medical history (e.g., duration of diabetes, medications), exercise history (i.e., Godin Leisure Time Exercise Questionnaire), as well as HbA1c, lipids in last 6 months and Creatinine within last year. We will also measure HbA1c with a point of care device (DCA vantage) which requires a single drop of blood (similar demands as a capillary glucose measurements that people with diabetes perform routinely). Body composition with be estimated with bioelectrical impedance analysis (BIA, Tanita TBF-300A). During this initial visit, participants will also have the opportunity to practice walking on a treadmill at the speed and grade that will be assigned during the intervention period (5.0km/hr at a grade of 0.5%).

Experimental Protocol: Walking Conditions and seated control conditions. Participants will complete standardized bouts of 50 minutes of walking at ~3.5 metabolic equivalents (METs), which is equivalent to 5.0 km/h at 0.5% incline. This is chosen to represent the typical physical activity prescription for prevention and treatment of T2D and its complications (i.e., 150 minutes per week of moderate activity [3-5.9 METs] performed over 3 days of the week). A standardized 5-minute warm-up and cool-down will be included at a pace of 3.5 km/h at 0% grade. If a participant cannot comfortably complete 15 minutes of walking at this intensity in the baseline screening visit they will be allowed to reduce the speed to 4.5 km/h (3.3 METs) or 4.0 km/h (3.1 METs) and this will be recorded. Heart rate and ratings of perceived exertion will be monitored during exercise and recorded every 10 minutes. Blood pressure and capillary blood glucose will be monitored before and after exercise. Participants will complete this walking protocol in the fasted state, 3-4 hours post lunch, and 30 minutes post dinner. In the seated control condition, participants will sit quietly and be allowed to read, work on a computer and/or watch a video for 60 minutes to match the time spent walking in the alternate intervention. At the beginning and end of each walking and sedentary control condition, participants will be ask to expire into a mouth piece connected to a metabolic cart for the measurement of oxygen consumption and carbon dioxide production. With guidance from the study coordinator, participants will also perform a 24 hour recall of the foods they consumed on the previous day.

Standardized Diet: Participants will be provided with all their food (breakfast, lunch, dinner, and snacks) for two days in each condition. Macronutrient profile will be based on Diabetes Canada guidelines with meal/snack providing ~55% carbohydrate (focusing on low glycemic index), ~30% fat, and ~15% protein. Participants will be provided with a food log with prescribed timing for each meal and will be asked to complete this log to confirm compliance and record any deviations with the diet.

Summary of laboratory visits:

* Day 1. Participants will arrive to PADL at their designated appointment time and an individual will insert both the Medtronic and Freestyle Libre CGM. They will be given standardized meals at this visit which will be consumed on days 2 and 3.
* Day 2. Participants will arrive at PADL for the first of the 4 conditions. The randomization process will determine which of the conditions will be completed and the state (fasted or fed) that the participant will come in.
* Day 3. Standardized meals (breakfast, lunch, and dinner) will be consumed on day 3. There is no lab visit on day 3.
* Day 4. As a wash out day, participants will resume their typical daily activities and eating habits which will be recorded in their log books.
* Day 5. Participants will complete condition 2 on this day. Standardized meals will be consumed.
* Day 6. Standardized meals (breakfast, lunch, and dinner) will be consumed on day 6. There is no lab visit on day 3.
* Day 7.The Medtronic CGM will be taken out and replaced with another Medtronic device (Note: the Medtronic CGM lasts for 6 days while the newer Abbott CGM lasts for 14 days). Standardized meals will be consumed on this day.
* Day 8. Condition 3 will be completed on this day. Standardized meals will be consumed.
* Day 9. No lab visit this day. Standardized meals will be consumed.
* Day 10. As a wash out day, participants will resume their typical daily activities and eating habits which will be recorded in their log books.
* Day 11. Participants will complete condition 4 on this day. Standardized meals will be consumed.
* Day 12. Standardized meals (breakfast, lunch, and dinner) will be consumed on day 6 and then the CGMs will be removed.

Analyses. Data from both CGMs will be compared between the 24-hour periods which follow each intervention. Parameters of interest include post meal area under the glucose curve, mean glucose, glycemic variability, fasting glucose, time spent in hyperglycemia (>10mmol/l), and time spent in hypoglycemia (<4mmol/l). A one-way Anova will be used to compare the 4 conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D for more than 6 months
* 30-90 years of age
* Able to understand English or French and comply with study requirements (e.g., attend visits during the day)

Exclusion Criteria:

* Contraindications to exercise (PAR-Q+, Rose Angina questionnaire, limited ability to walk for 50 min).
* Allergies or dietary restriction that could prevent adherence to standardize meals.
* Previous myocardial infarction, stroke or diagnosed coronary artery disease
* Changes in diabetes medication in last 3 months
* Treated by insulin or corticosteroids
* Change in body weight (>5%) in last 3 months
* Blood pressure >160/100 mmHg; resting heart rate>100

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Mean 24-hour glucose | Within the 24 hours following exercise or control
  Glucose measured by continuous glucose monitoring over 24 hours starting at the beginning of exercise on seated control

SECONDARY OUTCOMES:
Postprandial glucose | Within the 24 hours following exercise or control
  The mean of the 2-hour glucose concentrations following breakfast, lunch and dinner
Glucose variability | Within the 24 hours following exercise or control
  Calculated as the mean amplitude of glycemic excursion (i.e. MAGE)
Fasting glucose | Within the 24 hours following exercise or control
  The mean of 3 consecutive continuous glucose monitoring values before breakfast
Energy expenditure (METs) | Within the 50 minutes of exercise or control
  This outcome is assessed by the metabolic cart during exercise
Respiratory Exchange Ratio (RER) | Within the 50 minutes of exercise or control
  This outcome is assessed by the metabolic cart during exercise

CONTACTS AND LOCATIONS:
Overall Officials: Normand Boule, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada